CLINICAL TRIAL: NCT02223598
Title: A Phase 1, Dose-Escalation/Dose-Expansion Study Evaluating the Safety, Pharmacokinetics and Pharmacodynamic Effects of Orally Administered CB-5083 in Subjects With Lymphoid Hematological Malignancies
Brief Title: A Phase 1 Study Evaluating CB-5083 in Subjects With Lymphoid Hematological Malignancies
Acronym: CLC-102
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: MTD determined
Sponsor: Cleave Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLC-102
Record Dates: First submitted 2014-08-15; First posted 2014-08-22 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2017-06

CONDITIONS: Lymphoid Hematological Malignancies; Relapsed and Refractory Multiple Myeloma
Keywords: Lymphoid Hematological Malignancies
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — CB-5083; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Escalation - CB-5083 (Experimental): CB-5083 will be administered orally, 4 days on and 3 days off, for 28 day cycles, as a single agent to subjects with lymphoid hematological malignancies
  Interventions: Drug: CB-5083
- Dose Expansion - CB-5083, Dexamethasone (Experimental): CB-5083 will be administered orally, 4 days on and 3 days off, for 28 day cycles, as a single agent to subjects with relapsed and refractory multiple myeloma; in addition, subjects who develop progressive disease at the end of Cycle 1, or beyond, may receive their current dose of CB-5083 in combination with oral or IV low dose Dexamethasone (40 mg)
  Interventions: Drug: CB-5083; Drug: Dexamethasone
- Dose Expansion - CB-5083 (Experimental): CB-5083 will be administered orally, daily, 4 days on and 3 days off, for 28 day cycles, as a single agent to subjects with diffuse large B-cell lymphoma (DLBCL) or Waldenstrom Macroglobulinemia, if such arm is opened, per Sponsor
  Interventions: Drug: CB-5083

INTERVENTIONS:
Drug: CB-5083
Drug: Dexamethasone
  Arms: Dose Expansion - CB-5083, Dexamethasone

SUMMARY:
The purpose of this study is to determine the safety, tolerability, dose limiting toxicities, and maximum tolerated dose of CB-5083 in subjects with lymphoid hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age at the time of signing the consent form.
2. Dose Escalation Phase: Have a documented diagnosis of a lymphoid hematological malignancy as described by the 2008 World Health Organization (WHO) classification that requires therapy and for which there is no standard of care or standard of care is not expected to be effective. Subjects must not be candidates for anti-tumor regimens known to provide clinical benefit.

   MM Dose Expansion Cohort:
3. Must have a documented diagnosis of relapsed and refractory multiple myeloma defined by the International Myeloma Working Group (IMWG) criteria.
4. Must have measurable disease defined as:

   * Serum M-protein ≥ 0.5g/dL of IgA or ≥ 1 g/dL of IgG, or
   * Urine M-protein ≥ 200 mg/24 hr, or
   * Involved FLC assay > 10 mg/dL with abnormal FLC ratio.
5. Must have received at least 4 prior therapies, including an alkylating agent (unless not clinically indicated), proteasome inhibitor, an immunomodulatory (IMiD) and CD38 targeted therapy. At least 3 prior therapies where CD38 targeted therapies are not approved, not commercially accessible, contraindicated or refused by subject.

   DLBCL Dose Expansion Arm:
6. Must have histologically confirmed DLBCL that is relapsed or refractory to previous therapy.
7. Must have ≥1 measurable disease sites as defined by standard Lugano classification.
8. Must have received at least 2 prior therapies, including a CD20 targeted therapy, alkylating agent or corticosteroid; subjects who are not eligible for high-dose chemotherapy and autologous stem cell transplantation (HD-ASCT) are eligible with exposure to at least 1 prior therapy.

   Waldstrom's Macroglobulinemia Dose Expansion Arm:
9. Must have a confirmed diagnosis of WM as defined by the Second International Workshop, with a clinical indication for treatment.
10. Must have measurable disease, defined as presence of serum immunoglobulin M (IgM) with a minimum IgM level of ≥ 2 times the upper limit of each institution's normal value is required.
11. Must have relapsed/refractory disease after receiving 1 or more lines of therapy, including a Bruton tyrosine kinase (BTK) inhibitor (eg ibrutinib) if approved by the local health authority and commercially accessible.

    All Arms:
12. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2.
13. Adequate bone marrow function without transfusion or growth factor support, defined as:

    * Absolute neutrophil count ≥ 1,000/μL;
    * Platelet count ≥ 50,000/μL;
    * Hemoglobin ≥ 8.0 g/dL
14. Adequate organ function defined as:

    * Serum creatinine ≤ 1.5 mg/dL or creatinine clearance > 45 mL/min according to Cockcroft-Gault formula; (If creatinine clearance calculated from a 24-hour urine sample is ≥45 mL/min, the subject will qualify for the study).
    * Serum total bilirubin ≤ 2.0 mg/dL (34.2 μmol/L); or > 3.0 × upper limit of normal (ULN) for subjects with hereditary benign hyperbilirubinemia
    * AST (SGOT) ≤ 3 × the ULN;
    * ALT (SGPT) ≤ 3 × the ULN;
15. Subjects who are fertile agree to use an effective barrier method of birth control (ie, latex condom, diaphragm, cervical cap, etc) to avoid pregnancy. Female subjects need a negative serum or urine pregnancy test within 7 days of study enrollment (applies only if subject is of childbearing potential. Non-childbearing is defined as ≥ 1 year postmenopausal or surgically sterilized).
16. Willing and able to provide written Informed Consent and adhere to study procedures.

Exclusion Criteria:

1. Subjects with leukemia are excluded, with the exception of chronic lymphocytic leukemia (CLL), who are allowed in the dose escalation phase. Subjects with Burkitt lymphoma, plasma cell leukemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes), or amyloidosis are also excluded.
2. Clinically active central nervous system (CNS) cancer involvement. Imaging to exclude CNS involvement not required.
3. Previous or concomitant malignancy, except for basal-cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the uterine cervix. Subjects with other malignancies are eligible if they have remained disease free for at least 2 years prior to study entry;
4. Use of any anti-cancer drug therapy within 14 days prior to Baseline (within 28 days for monoclonal antibodies [eg anti-CD38]).
5. Use of any investigational agent within 28 days prior to Baseline.
6. Presence of clinically significant non-hematological toxicity of prior chemotherapy that has not resolved to ≤ Grade 1 as determined by CTCAE v 4.0, with the exception of alopecia and peripheral neuropathy. Note: Peripheral neuropathy > Grade 2 plus pain, or Grade 3 or Grade 4 are excluded.
7. Radiotherapy within 14 days prior to Baseline.
8. Major surgery within 6 weeks prior to Baseline. The subject must have recovered from surgery and be without current complications of infection or dehiscence.
9. Peripheral autologous stem cell transplant within 12 weeks prior to Baseline; prior allogeneic transplants within 16 weeks or chronic use of immunosuppressants.
10. Active infection requiring systemic therapy, including known human immunodeficiency virus (HIV), acquired immunodeficiency syndrome-related illness, or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
11. Major cardiac abnormalities as defined but not limited to the following: uncontrolled angina or unstable life-threatening arrhythmias, history of myocardial infarction within 12 weeks prior to Baseline, Class 3 or higher New York Heart Association (NYHA) congestive heart failure, or severe cardiac insufficiency, persistent (3 consecutive electrocardiograms (ECGs) performed ≥ 5 minutes apart) prolongation of the QTc (Fridericia) interval to > 480 msec.
12. Cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 12 weeks prior to Baseline.
13. Major gastrointestinal (GI) disease as defined but not limited to the following: history of inflammatory bowel disease or other illness resulting in chronic diarrhea, known achlorhydria or history of GI surgery that could reduce the acidity of the stomach, acute pancreatitis or cholecystitis within 6 months prior to Baseline, or GI disease that may interfere with the absorption of orally-administered drugs.
14. Grade 3 or 4 eye disorder at study entry, unless stable and longstanding (>3 months) and unlikely to interfere with protocol-required ophthalmology assessments.
15. A condition that is expected to require concomitant use of any medication listed as prohibited while on study.
16. Is a pregnant or lactating female.
17. Has any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of the study results and, in the Investigator's opinion, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-08-25 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicities (DLTs) of oral CB-5083 in subjects with lymphoid hematological malignancies | Dose Escalation Stage - the first 28 days of treatment (Cycle 1) with CB-5083
To determine the pharmacokinetic (PK) profile of oral CB-5083 in subjects with lymphoid hematological malignancies by measuring the AUC | Dose Escalation and Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 in the second 28 days (Cycle 2) of treatment with CB-5083
To determine the PK profile of oral CB-5083 in subjects with lymphoid hematological malignancies by measuring the Cmax | Dose Escalation and Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 of Cycle 2 of treatment with CB-5083
To determine the PK profile of oral CB-5083 in subjects with lymphoid hematological malignancies by measuring the Cmin | Dose Escalation and Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 of Cycle 2 of treatment with CB-5083
To determine the PK profile of oral CB-5083 in subjects with lymphoid hematological malignancies by measuring the Tmax | Dose Escalation and Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 of Cycle 2 of treatment with CB-5083
To determine the PK profile of oral CB-5083 in subjects with lymphoid hematological malignancies by measuring the T1/2 | Dose Escalation and Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 of Cycle 2 of treatment with CB-5083
To confirm the safety and tolerability of oral CB-5083 administered to subjects with relapsed and refractory Multiple Myeloma at the maximum tolerated dose (MTD) at the end of the Dose Escalation Stage | Dose Expansion Stage - from day 1 of Cycle 1 through 28 days after the patient's last cycle of treatment
To confirm the safety and tolerability of oral CB-5083 administered to subjects with relapsed/refractory DLBCL or Waldenstrom Macroglobulinemia at the MTD | Dose Expansion Stage - from day 1 of Cycle 1 through 28 days after the patient's last cycle of treatment

SECONDARY OUTCOMES:
To assess the pharmacodynamic (PD) effects of CB-5083 in peripheral blood cells and cancer cells | Dose Escalation and Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1
To further asses the PK profile of oral CB-5083 in subjects by measuring the AUC | Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 of Cycle 2 of treatment with CB-5083
To further asses the PK profile of oral CB-5083 in subjects by measuring the Cmax | Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 of Cycle 2 of treatment with CB-5083
To further asses the PK profile of oral CB-5083 in subjects by measuring the Cmin | Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 of Cycle 2 of treatment with CB-5083
To further asses the PK profile of oral CB-5083 in subjects by measuring the Tmax | Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 of Cycle 2 of treatment with CB-5083
To further asses the PK profile of oral CB-5083 in subjects by measuring the T1/2 | Dose Expansion Stages - days 1, 2, 4 and 5 of Cycle 1 and days 1 and 2 of Cycle 2 of treatment with CB-5083
To evaluate preliminary efficacy of oral CB-5083 in subjects, using standard response criteria | Dose Expansion Stages - at the end of each 28 day cycle of treatment

OTHER OUTCOMES:
To assess the predictive value of potential baseline biomarkers for clinical trial subject enrichment strategies | Dose Expansion Stages - within 28 days before day 1 of Cycle 1

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - RCCA MD, Bethesda, Maryland
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Cedars Cancer Centre, McGill University Health Centre, Montreal, Quebec